CLINICAL TRIAL: NCT02106481
Title: Comparison of a Single Shot Femoral Nerve Block to Femoral Nerve Block Shot Plus Continuous Femoral Nerve Catheter for Total Knee Replacement Surgery; a Randomized, Blinded Controlled Trial.
Brief Title: Comparing Femoral Nerve Catheters to Single Shot Femoral Nerve Blocks for Total Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Maine Medical Center (Other)
Responsible Party: Principal Investigator, Varun Dixit, Anesthesiologist, Eastern Maine Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-1-M-255
Record Dates: First submitted 2014-03-27; First posted 2014-04-08 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Knee Osteoarthritis
Keywords: TKA; TKR; Knee OA; pain management; Femoral Nerve Catheter; Single Shot Femoral Nerve Blocks
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoral Nerve Catheters (Active Comparator): Patients will receive a Single Shot Femoral Nerve Block along with a conventional continuous femoral nerve catheter
  Interventions: Drug: Femoral Nerve Catheters; Drug: Single Shot Femoral Nerve Blocks
- Single Shot Femoral Nerve Blocks (Active Comparator): Patients will receive a Single Shot Femoral Nerve Block and a sham catheter post op.
  Interventions: Drug: Single Shot Femoral Nerve Blocks

INTERVENTIONS:
Drug: Femoral Nerve Catheters — Catheter will be bolused with 0.5 % ropivacaine around the femoral nerve and occlusive dressing applied over the catheter.
  Patients with CFNB will receive ropivacaine 0.2% infusion (the infusion rate will be dependent on the clinical judgement of the anaesthesiologist)
  Other Names: 0.5% ropivacaine bolus followed by 0.2% infusion
  Arms: Femoral Nerve Catheters
Drug: Single Shot Femoral Nerve Blocks — The group with SSFNB will receive a femoral nerve block before the surgery in the pre-operative area guided by a nerve stimulator and ultrasound. A bolus of 0.5 % ropivacaine will be injected around the femoral nerve.
  Other Names: 0.5% ropivacaine

SUMMARY:
The purpose of this study is to compare two methods of pain control used during total knee joint replacement surgery. The pain medication that will be used for this study is not experimental.

The investigators will compare the single shot femoral nerve block (SSFNB) and Femoral Nerve Block (FNB) plus continuous femoral nerve catheter (CFNC) to determine which method gives patients better pain control, increasing the capability to participate in physical therapy and decreasing the consumption of other pain medication. With either the single shot or the catheter the local numbing medication called ropivacaine will be used.

DETAILED DESCRIPTION:
The study will be a randomized controlled blinded study with a sham control arm. The patients will be randomized to either a single shot FNB with placement of a catheter on the skin (sham control) or a conventional CFNC with catheter.

The group with SSFNB will receive a femoral nerve block before the surgery in the pre-operative area guided by a nerve stimulator and ultrasound. A bolus of 0.5 % ropivacaine will be injected around the femoral nerve. A catheter would be placed on the skin, without penetration, with occlusive dressing applied over the site. A standard size saline bag will be placed on the pump but will not be turned on. The tubing will be opaque and a bag will be placed over the pump to blind the patient to the medication, or lack of medication, being administered. The patient, nursing staff and physical therapists will be blinded to the presence of a sham catheter. The infusion will be labelled 'Study Drug R' or 'Study Drug N' in the electronic medicine prescription.

The group randomized with active drug by CFNB would have a continuous femoral catheter placed using nerve stimulator and ultrasound. Catheter will be bolused with 0.5 % ropivacaine around the femoral nerve and occlusive dressing applied over the catheter.

After placement of the femoral nerve block patients will be transported to the operating room and spinal anesthesia with bupivacaine and fentanyl will be performed. Intra-operative sedation of propofol infusion will be titrated to the discretion of the anaesthesia team. Patients will receive scheduled as well as rescue analgesia as per clinical pathway protocol.

Patients with CFNB will receive ropivacaine 0.2% infusion (the infusion rate will be dependent on the clinical judgement of the anaesthesiologist) in the post anaesthesia care unit (PACU) after the spinal anaesthesia has worn off. The infusion will be continued for the duration of the catheter, 4am POD one. Patients with SSFNB will not receive any infusion through the sham catheter.

The catheters will be removed on post-operative day (POD) one at about 8 am. Patient's pain score using visual analogue score (VAS) will be assessed. Functional status will be assessed by the physical therapist on POD one. The therapist will assess and document the distance walked, assistive device used, level of assist needed to ambulate, and knee proprioception or continued recommendation of the knee immobilizer.

Patients will be assessed in the PACU and POD 1 and 2. Recordings will be made of total opioid consumption in morphine equivalents, VAS score from 0-10 both at rest and on participation in physical therapy, incidence of nausea and vomiting and functional status during physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-80 years old)
* Scheduled to undergo primary unilateral TKA with Parapatellar approach
* Patient agrees to participate in the study
* Effective femoral nerve block
* No contraindication for spinal or regional anesthesia

Exclusion Criteria:

* History of opioid dependence or current chronic analgesic therapy (daily use >4 weeks
* Allergy to study medications
* Known hepatic or renal insufficiency/disease
* Peripheral neuropathy
* Morbid obesity (BMI >40 kg/m2)
* Unable to comply with study protocol
* Pregnancy
* Incarceration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain | 48 hours post operatively
  Pain Analog Scale- 0-10 were 10 is the worst possible pain and 0 is no pain at all.

OTHER OUTCOMES:
Restfulness of sleep | 8 AM post op day 1
  Patients will be asked if they had difficulty sleeping because of pain.
Nausea and Vomiting | 8 AM post op day 1
  Nausea and Vomiting- Written questionnaire administer to patient. Did the patient experience Nausea? Yes/No. Using scale 0- no nausea, 1- nausea no vomiting, 2-vomiting, 3- persistent vomiting.
Distance Walked | 8 AM post op day 1, 48 hours post op, 3 months post op
  Distance walked- Distance will be measured in meters and assistive device used (including knee immobilizer)
Level of Assist for Ambulation | 8 AM post op day 1, 48 hours post op, 3 months post op
  Level of Assist for Ambulation- Independent (no device, timely, safely), modified independent (assistive device, safely or timeliness issues) supervision (requires standby assist, cueing), minimal assist (patient expends 75% of effort needed to completed task) , moderate assist (patient expends 50-74% of effort needed to completed task), max assist (patient expends 25-49% of effort needed to completed task), total assist (patient expends >25% of the effort needed to complete task).
Hours until knee immobilizer is discharged | 8 AM post op day 1, 48 hours post op, 3 months post op
  Hours until knee immobilizer is discharged - As a gauge of knee proprioception and quad strength the physical therapist will discharge the knee immobilizer when the patient can safely mobilize without the brace. The hours from surgery to discharge will be measured and >24 hours after surgery will be considered delayed discharge where <24 hours post op will be considered satisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Varun Dixit, MD, Principal Investigator — Eastern Maine Medical Center
Locations (1):
- Eastern Maine Medical Center, Bangor, Maine, United States